CLINICAL TRIAL: NCT03772236
Title: Evaluation of the Relation Between the Rotation Angle of the Talar Component and the Antero-medial Pain in Patients Underwent Total Ankle Replacement, at Least One Year After Surgery
Brief Title: Phi Angle and Antero-medial Pain in Total Ankle Replacement Follow-up
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: ARP2
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Ankle Osteoarthritis; Prostheses and Implants
Keywords: Total Ankle Replacement; Pain Measurement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study evaluates the relation between the rotational alignment of the talar component (phi angle) and the antero-medial ankle pain in patients underwent total ankle replacement, at least one year after surgery.

Moreover, the study aims to define a range of the phi angle associated with a lower frequency of antero-medial pain.

DETAILED DESCRIPTION:
Background:

In case of total ankle prosthesis surgery, the correct positioning of the talar component is one of the most challenging tasks. When performing total ankle replacement, the primary goal for long-term implant survival is to restore a physiological alignment of the prosthesis in the lateral and frontal planes. In fact, an incorrect alignment can alter joint mechanics and joint reactive forces that can lead to implant failure (Saltzman, 2004).

Regarding the rotation in the dorsoplantar plane, the prosthesis is aligned taking as reference the axis of the second metatarsal bone, with the foot in neutral position (Roukis, 2015). In this regard, there are no specific mechanical-articular considerations as for the lateral and frontal planes. However, it is expected that misalignments of the prosthesis in the dorsoplantar plane may involve the presence of antero-medial pain in the ankle in the long term (at least 1 year after surgery).

At present, no previous studies have verified whether there is a relation between the rotational alignment of the talar component in the dorsoplantar plane and the frequency of antero-medial ankle pain, at least 1 year after surgery. This evaluation can provide useful information for a more advantageous placement of the implant during the intervention.

Aim of the Study:

The aim of the study is to evaluate the relation between the rotational alignment of the talar component (phi angle) and the antero-medial ankle pain, in patients underwent total ankle replacement, at least one year after surgery.

Moreover, the study aims to define a range of the phi angle associated with a lower frequency of the antero-medial pain.

Methods:

A sample of 100 subjects in the follow-up period after total ankle replacement (minimum 12 months after surgery, maximum 36 months) will be enrolled. Age range will be 18 to 60 years. Each subject will be evaluated once, in occasion of the routine follow-up examination. The subjects will be enrolled consecutively and differentiated according to the time passed since the intervention (at least 12 months), with incremental windows of 6 months, up to a maximum of 36 months. This will lead to define 4 time windows (12-18 months, 18-24, 24-30, 30-36). A number of 25 subjects will be enrolled for each time window. Once a time window will be completed, only subjects belonging to the remaining not completed windows will be enrolled.

Outcomes:

The phi angle will be measured according to that described by Manzi et al., 2017. Specifically, the phi angle will be obtained by the orthopaedist on the standard dorsoplantar radiograph of the foot, which is routinely performed for the follow-up examination. The phi angle is the relative angle between the alignment of the talar component of the implant, and the axis passing through the second metatarsal bone, in the dorsoplantar plane. The phi angle is defined as negative when the talar component is aligned in an abducted position to the second metatarsal axis; similarly, the angle is defined as positive when the talar component is aligned in an adducted position.

The rate of postoperative pain will be assessed during the follow-up examination by a recently distributed pain monitoring web-based app: 'NavigatePain' (NavigatePain, Aglance Solutions, Denmark). The app is used in a simple and intuitive manner by exploiting tablet device (Boudreau, 2016; Matthews, 2018). It is used only for data collection, without therapeutic or diagnostic purposes. In few minutes, it allows the patient to draw the pain areas in the frontal and lateral planes, automatically providing an index that quantifies the percentage of anterior and medial areas affected by pain (with respect to the whole body area in the considered plane).

The antero-medial ankle pain will be obtain as the sum of the anterior and medial pain indexes provided by the app.

The strength of the relation between the phi angle and the antero-medial ankle pain will be evaluated according to Pearson correlation coefficient, or Spearman rank correlation in case of not normal distribution. Statistical significance of the coefficients will be tested according to two-tailed t-test or permutation distribution test assessing Pearson and Spearman coefficients, respectively. Linear regression analysis will be performed as well.

Correlation coefficient and linear regression will be evaluated in each time window. The results will be compared among the consecutive windows in order to assess the potential dependence on the follow-up time.

The sample size of 25 subjects per time window has been verified to guarantee identifying as significantly different from zero a correlation value larger than 0.7 (i.e. strong correlation), by t-test at 0.05 level alpha and power 95% (G*Power software, Universitat Dusseldorf, Germany).

The distribution of the pain rate will be evaluated in function of the phi angle. Potential threshold values of phi associated with lower pain rates will be identified, in order to define a range of phi associated with a lower frequency of the antero-medial pain.

ELIGIBILITY:
Inclusion Criteria:

* previous intervention of first implant of total ankle replacement, with at least 12 months of follow up and maximum 36 months

Exclusion Criteria:

* more than 36 months from the surgery of first implant of total ankle replacement
* previous revision surgery of ankle prosthesis
* previous intervention of ankle disarthrodesis and ankle prosthesis implant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing follow-up examination at a third-level hospital after total ankle replacement
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Phi angle | Through study completion, an average of 18 months
  Relative angle (measured in degrees) between the alignment of the talar component of the implant, and the axis passing through the second metatarsal bone, in the dorsoplantar plane.
Antero-medial ankle pain | Through study completion, an average of 18 months
  Sum of the antero and medial pain areas, measured as percentage with respect to the total body area in the considered plane.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Usuelli, MD, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- Irccs Istituto Ortopedico Galeazzi, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boudreau SA, Badsberg S, Christensen SW, Egsgaard LL. Digital Pain Drawings: Assessing Touch-Screen Technology and 3D Body Schemas. Clin J Pain. 2016 Feb;32(2):139-45. doi: 10.1097/AJP.0000000000000230. PMID 25756558
- [Background] Manzi L, Villafane JH, Indino C, Tamini J, Berjano P, Usuelli FG. Reliability of the Phi angle to assess rotational alignment of the talar component in total ankle replacement. Foot Ankle Surg. 2019 Apr;25(2):169-173. doi: 10.1016/j.fas.2017.10.009. Epub 2017 Nov 8. PMID 29409284
- [Background] Matthews M, Rathleff MS, Vicenzino B, Boudreau SA. Capturing patient-reported area of knee pain: a concurrent validity study using digital technology in patients with patellofemoral pain. PeerJ. 2018 Mar 8;6:e4406. doi: 10.7717/peerj.4406. eCollection 2018. PMID 29568700
- [Background] Roukis TS. The Salto Talaris XT Revision Ankle Prosthesis. Clin Podiatr Med Surg. 2015 Oct;32(4):551-67. doi: 10.1016/j.cpm.2015.06.019. Epub 2015 Jul 31. PMID 26407741
- [Background] Saltzman CL, Tochigi Y, Rudert MJ, McIff TE, Brown TD. The effect of agility ankle prosthesis misalignment on the peri-ankle ligaments. Clin Orthop Relat Res. 2004 Jul;(424):137-42. doi: 10.1097/01.blo.0000132463.80467.65. PMID 15241155